CLINICAL TRIAL: NCT01643759
Title: A Single Dose PK Study of BTDS 5, 10, and 20 in Chinese Osteoarthritis Patients
Brief Title: Norspan Transdermal Patches Study in Osteoarthritis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP08-CN-002
Record Dates: First submitted 2011-11-17; First posted 2012-07-18 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Osteoarthritis Disorders
Keywords: osteoarthritis disorders
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- buprenorphine transdermal system (Experimental): buprenorphine transdermal system
  Interventions: Drug: buprenorphine

INTERVENTIONS:
Drug: buprenorphine — The subjects will be randomized to receive either a single dose of BTDS 5, or BTDS 10, or BTDS 20 for 7 days. Plasma concentrations of buprenorphine and norbuprenorphine will be analyzed to determine the following pharmacokinetic parameters: AUC0-t:pg•hr/ml-Area under the plasma concentration-time curve frame: predose,6,12,24,36,48,60,72,96,120,144,168,169,170,171,172,174,180,192,216,240 hours post-dose.AUC0-inf:pg•hr/ml-Area under the plasma concentration-time curve extrapolated to infinity. Cmax: pg/ml-Maximum observed plasma buprenorphine concentration. Tmax: hrs-time at which Cmax is first observed. t½: Apparent half life of buprenorphine elimination.
  Other Names: Norspan

SUMMARY:
This is a single center, open label, randomized, parallel group single dose pharmacokinetic (PK) study.

DETAILED DESCRIPTION:
After up to 7-day screening period, Eligible Patients will be randomized to 1 of 3 treatment groups, and begin treatment with BTDS 5mg, 10mg,20mg for 7 days.Venous blood will be collected at 0, 6, 12, 24, 36, 48, 60, 72, 96,120, 144,168,169,170,171,172,174,180,192,216, 240 h postdose respectively.Plasma concentrations of buprenorphine and norbuprenorphine will be analyzed to determine the following pharmacokinetic parameters: AUC0-t, AUC0-inf, Cmax, Tmax, t½.

ELIGIBILITY:
Inclusion Criteria:

* Patients volunteering for participation in the study.
* Male and female patients with diagnosis of osteoarthritis, age from 20 to 60 years.
* Body weight ≥ 50kg , and BMI range ≧ 18.5, ﹤ 30.
* Having the results within the following ranges and having been judged as eligible for the study participation by the investigator:Systolic blood pressure (supine), 90-140 mm Hg,Diastolic blood pressure (supine), 60-90 mm Hg, Armpit body temperature, 35.0-37.5 degree Celsius.
* Agreed not to use any medication (except vitamins or mineral supplements) during the course of the study.
* Have not smoked or chewed tobacco for at least 45 days prior to dosing with study drugs, and agree not to use tobacco products during the study.
* Females of childbearing potential must have a negative serum pregnancy test during screening visit and at check-in.

Exclusion Criteria:

* Subjects who have been taking opioid analgesic formulations excess 7 days within 3 months of Visit 1.
* Subjects who have been taking CYP3A4 inhibitor or inducer within the last 1 month prior to the screening visit.
* Subjects who have been taking any medication including OTC (except vitamin and/or mineral supplements) within 7 days prior to the first dose of the trial product.
* Patients who have a current chronic disease(s), or who have a past history and high possibilities to relapse, in addition to their musculo-skeletal pain, requiring frequent analgesic therapy.
* Subjects with clinically unstable respiratory disease, dysfunction of the biliary tract, thyroid disease, adrenal cortical insufficiency, prostatic hypertrophy requiring intervention or renal artery stenosis.
* Subject who have a past history of malignant neoplasm.
* Subjects with clinically unstable, active or symptomatic heart disease.
* Subjects who have psychiatric disorder, uncontrolled seizures or convulsive disorder and so on.
* Subjects who have any medical or surgical conditions that might interfere with transdermal absorption, distribution, metabolism, or excretion of drugs.
* History of frequent nausea or emesis regardless of etiology.
* Subjects who have a current or past history of substance or alcohol abuse, or subjects who give a positive result in drug abuse test during the Screening Period.
* Subjects scheduled for therapies within the study period which might effect study assessment.
* Subjects with values > 2 times the upper limit of normal for AST or ALT or total bilirubin during the Screening Period or who have severe impaired liver function.
* Subjects with serum creatinine > 2 mg/dL during the Screening Period or who have severe impaired renal function.
* Subjects with serum potassium < 3.5 mEq/L during the Screening Period.
* Subjects with positive result of anti-human immunodeficiency virus antibodies, hepatitis B surface antigen, hepatitis C virus antibody or qualitative syphilis tests.
* Donated 400 mL or more of blood or blood products within 3 months prior to the start of the study, or donated 200 mL or more of blood or blood products within 1 month prior to the start of the study.
* Subjects who have a history of supersensitivity to study drug.
* Subjects who participated in a clinical research study within 1 month of study entry.
* Subjects who participated previously in a BTDS study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Pre-dose, 6hr, 12hr, 24hr, 36hr, 48hr, 60hr, 72hr, 96hr, 120hr, 144hr,168hr, 169hr, 170hr, 171hr, 172hr, 174hr, 180hr, 192hr, 216hr, 240hr post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Mundipharma China Ltd., Study Chair — Mundipharma China Ltd.
Locations (1):
- Investigational Site: Peking Union Medical Hospital(PUMC), Beijing, China